CLINICAL TRIAL: NCT03764852
Title: Feasibility Study on Laparoscopic Double-mesh Sacrocolpopexy With or Without Robotic Assistance, in Female Patients Presenting With Symptomatic Pelvic Organ Prolapse, Based on an Outpatient Treatment Model.
Brief Title: AMBULAPSE STUDY Feasibility Study on Laparoscopic Double-mesh Sacrocolpopexy With or Without Robotic Assistance, in Female Patients Presenting With Symptomatic Pelvic Organ Prolapse, Based on an Outpatient Treatment Model.
Acronym: AMBULAPSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-PP-12
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Pelvic Organ Prolapse
Keywords: outpatient
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- outpatient laparoscopic (Experimental): Patients will have laparoscopic outpatients. The procedure is identical to that performed in hospital. What changes is that the patient will return home at night if her condition allows it.
  Interventions: Procedure: outpatient laparoscopic

INTERVENTIONS:
Procedure: outpatient laparoscopic — The intervention is a outpatient laparoscopic sacrocolpopexy with robotic assistance.
Procedure: outpatient laparoscopic — The intervention is a outpatient laparoscopic sacrocolpopexy without robotic assistance.

SUMMARY:
Pelvic organ prolapse is an increasingly common functional disorder which affects approximately 30 to 40% of the female population, 12% of whom have a symptomatic form, with a psychological, physical and social impact. Laparoscopic sacrocolpopexy represents the surgical "gold standard" for the treatment of this functional disorder. It aims to suspend the vaginal vault by means of a prosthesis. The patient satisfaction rate is evaluated at 94% with low overall complication rate, evaluated at 11%.

Pelvic organ prolapse surgery is a common, with an estimated 30,000 procedures carried out in France in 2013 (excluding hysterectomy) (2013 ATIH data), and the number will increase in the future due to increasing life expectancy. 13% of women will undergo this type of procedure. The French General Directorate of Health Care Supply (DGOS) deems outpatient surgery to be the benchmark for surgical activity in all eligible patients, and has expressed the need for recommendations and tools for supporting its development. The rate of outpatient surgery for prolapse remains low in France (6.1%, 2015 ATIH data), while it is 25% in the US and 56% in Denmark. The average duration of hospital stays for DRG N81.2 (first degree uterine prolapse) in 2015 was 3.43 days. These procedures have been the subject of publications concerning outpatient care and involving low numbers of patients, with the exception of the publication by Sinhal which involved 111 patients.

DETAILED DESCRIPTION:
In our study, the investigators propose to evaluate the success rate for outpatient laparoscopic sacrocolpopexy with or without robotic assistance in screened patients. With this aim in mind, the investigators will conduct a national multicenter prospective study including 80 female patients. Successful outpatient treatment is defined by the absence of conventional inpatient admission with 24H after surgery, the indications for admission being a CHUNG Score < 9, one perioperative complication, postoperative urinary retention requiring reinsertion of a urinary catheter. The outpatient success rate for other surgical techniques such as cholecystectomy or laparoscopic hysterectomy is above 90% in the literature. Envisaging an equivalent rate after laparoscopic sacrocolpopexy, our population size would make it possible to obtain precision +/- 5.3% for estimation of this proportion. The patients are followed up for 1 month with a postoperative visit at 30 days, during which the efficacy of the technique is evaluated using conventional indicators (POP-Q; ICIQ, USP, PFDI-20, PISQ-12, PFIQ-7, etc.). Once completed, this preliminary investigation will make it possible to define a reference value for successful outpatient sacrocolpopexy, which has not yet been published, which may be used as a basis for a larger scale randomized study that would aim to compare the efficacy of outpatient treatment, with conventional inpatient treatment, for efficient patient management

ELIGIBILITY:
Inclusion Criteria:

* woman between 40 and 80 years old
* Patient with significant prolapse POP-Q ≥ 2
* BMI <30
* ASA score ≤ 2
* sterile ECBU

Exclusion Criteria:

* Criteria related to the pathology or the organ:

  * History of pelvic cancer surgery
  * History of prolapse surgery
  * History of pelvic irradiation
  * Laying a concomitant urethral strip
  * Cervico-vaginal smear test not up to date.
  * Patient pregnant or having a desire for pregnancy
* Criteria related to concomitant treatments:

  * Cefazoline allergy
  * Taking the following medications within 48 hours
* Plavix®
* Vitamin K / Low Molecular Weight Healing Heparin

  * Contraindication to ambulatory care for medical reasons
* Sleep apnea syndrome
* Cardiopulmonary pathology
* Psychiatric pathology
* Hemorrhagic risk
* Diabetes imbalanced
* Unbalanced Hypertension

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only woman with pelvic organ prolapse
Enrollment: 80 (Estimated)
Dates: Start 2019-12-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Successful outpatient treatment | 24 hours after surgery
  Successful outpatient treatment is defined by the absence of conventional inpatient admission with 24H after surgery, the indications for admission being a CHUNG Score < 9, one perioperative complication, postoperative urinary retention requiring reinsertion of a urinary catheter

SECONDARY OUTCOMES:
The percentage of failure of the outpatient | 24 hours after surgery
  The percentage of failure of the outpatient is defined by the number of patients with a CHUNG score <9 in the outpatient department that does not allow the discharge of the patient or her admission to conventional hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Brannwel TIBI, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (5):
- France (5):
  - Hopital Antoine Beclere - Aphp, Clamart
  - Chu de Nantes, Nantes
  - CHU DE Nice - Hôpital l'Archet, Nice
  - Ch Lyon Sud, Pierre-Bénite
  - Hopital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drapier E, De Poncheville L, Dannappel T, Clerc P, Smirnoff A. [Day case laparoscopic sacral colpopexy for genital prolapse]. Prog Urol. 2014 Jan;24(1):51-6. doi: 10.1016/j.purol.2013.07.007. Epub 2013 Aug 13. French. PMID 24365629
- [Background] Bump RC, Norton PA. Epidemiology and natural history of pelvic floor dysfunction. Obstet Gynecol Clin North Am. 1998 Dec;25(4):723-46. doi: 10.1016/s0889-8545(05)70039-5. PMID 9921553
- [Result] Flam F. Sedation and local anaesthesia for vaginal pelvic floor repair of genital prolapse using mesh. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Dec;18(12):1471-5. doi: 10.1007/s00192-007-0350-8. Epub 2007 Mar 17. PMID 17370026
- [Result] Cuvelier G. [The ambulatory surgery, source of publications]. Prog Urol. 2013 Jun;23(7):427-9. doi: 10.1016/j.purol.2013.02.007. Epub 2013 Mar 26. No abstract available. French. PMID 23721700